CLINICAL TRIAL: NCT04053257
Title: Effect of Video Camera Monitoring Feedback on Hand Hygiene Compliance and Healthcare Associated Infections in Neonatal Intensive Care Unit, an Interventional Study
Brief Title: Effect of Video Camera Monitoring Feedback on Hand Hygiene Compliance and Infections in NICU
Acronym: CaM-HAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 09.2019.710
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Healthcare Associated Infection; Hand Hygiene; Neonatal Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Quasiexperimental, before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before intervention (No Intervention): HH opportunities, compliant moments and HAIs recorded before the intervention
- After intervention (Active Comparator): HH opportunities, compliant moments and HAIs recorded after the intervention
  Interventions: Other: Hand hygiene compliance observation with video camera surveillance system and performance feedback of the HH rates to HCWs

INTERVENTIONS:
Other: Hand hygiene compliance observation with video camera surveillance system and performance feedback of the HH rates to HCWs — Intervention:
  We will report baseline HH compliance rates and HAI rates to HCWs during a meeting where all HCWs are present. During this meeting we will remind major infection control measures, give examples of common mistakes they made without violating personal privacy rights of HCWs and patients.
  Arms: After intervention

SUMMARY:
The purpose of this study is to determine if use of the video camera surveillance system for HH observation and performance feedback about HH compliance rates can improve the HH compliance of HCWs and reduce healthcare-associated infections in the NICU.

DETAILED DESCRIPTION:
Hypothesis:

H1: Hand hygiene (HH) compliance monitoring using video camera surveillance and giving feedback of HH compliance rates to HCWs would effect the hand hygiene behavior of health care workers (HCW) and healthcare-associated infections (HAI).

Study design:

A video camera surveillance system is in place in all NICU rooms since 2018. The investigators designed a quasiexperimental (before-after) study.

Study site and participants:

The research will take place in NICU from July 2019 to March 2020. All nurses, attending physicians, resident physicians, environmental services staff, medical assistants work in NICU.

Control period (Before intervention):

We will observe HH behavior of HCWs using the video camera surveillance for four weeks. This will give us the baseline HH compliance rates of NICU.

The baseline HAI rates will be calculated of the 3 months before intervention.

Intervention:

We will report baseline HH compliance rates and HAI rates to HCWs during a meeting where all HCWs are present. During this meeting we will remind major infection control measures, give examples of common mistakes they made without violating personal privacy rights of HCWs and patients.

Experimental period (After intervention):

The investigators will perform HH observation for four weeks after the intervention. At the end of the observation period, feedback about the HH compliance rates, change and detailed analysis of HH compliance rates by indication, day of week, hour of the day and NICU rooms will be given during a second meeting with HCWs.

HAI rates will be calculated for period of 3 months after intervention.

Sustainability of the intervention:

We will measure HH compliance rates 12 weeks after the intervention to investigate the sustainability of our intervention.

A third meeting will be done with HCWs in the unit which the investigator give feedback about the HH compliance, HAI rates before and after the intervention periods.

Data collection:

Seven, trained HH observers will participate in the study. These observers will achieve at least 80% concordance before the study. HH compliance data will be collected using a mobile app. HH monitoring will be performed Monday through Sunday making observations from randomly selected 20 minutes lapses of morning (08:00 am - 04:59 pm), afternoon (05:00 pm - 11:59 pm) and night (00:00 am - 07:59 am) shifts of the day. All HCWs in the room during the 20 minutes observation period are monitored for HH opportunities. Each HH opportunity was stratified as compliant or noncompliant and was classified according to the three of WHO's My 5 Moments for HH as follows: (1) before touching a patient, (4) after touching a patient, and (5) after contact with the patient's environment. HH moments before an aseptic task (2) and after body fluid exposure risk (3) was not included due to low resolution of video camera surveillance system.

Compliance was calculated by dividing the total HH opportunities for each subject by the number of HH compliance × 100. Adequate materials for HH are defined using either the soap and water or alcohol-based handrub solution.

HAIs are identified and recorded by active surveillance method in NICU. HAIs are identified using CDC criteria.

Sample Size:

We used G-power program for sample size calculation. With a power of 90%, 0.05 type I error rate and anticipated HH compliance increase before and after intervention period as 10% we planned to record 538 HH opportunities for each period (1076 HH opportunities total)

ELIGIBILITY:
Inclusion Criteria:

- All HCWs working in the NICU during the study period.

Exclusion Criteria:

- Visiting patient relatives in the NICU during the study period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8335 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Total hand hygiene compliance of health care workers | 4 weeks
  By dividing the total HH opportunities for each subject by the number of HH compliance × 100
Health care associated infection rate | 12 weeks
  HAI number divided by the patient days in the unit

SECONDARY OUTCOMES:
Number of HH opportunities per minute | 4 weeks
  Total number of HH opportunities divided by total HH observation minutes
Hand hygiene compliance by indication | 4 weeks
  Dividing HH opportunities for each indication by HH compliance for each indication.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)